CLINICAL TRIAL: NCT02544633
Title: Phase 2, Parallel-Arm Study of MGCD265 in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With Activating Genetic Alterations in Mesenchymal-Epithelial Transition Factor
Brief Title: Phase 2 Study of MGCD265 in Patients With Non-Small Cell Lung Cancer With Activating Genetic Alterations in MET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 265-109
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Results first posted 2019-09-10 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Mirati; MGCD265; MET; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): MGCD265 in patients with MET activating mutations in tumor tissue
  Interventions: Drug: MGCD265
- Arm 2 (Experimental): MGCD265 in patients with MET gene amplifications in tumor tissue
  Interventions: Drug: MGCD265
- Arm 3 (Experimental): MGCD265 in patients with MET activating mutations in blood (circulating tumor DNA)
  Interventions: Drug: MGCD265
- Arm 4 (Experimental): MGCD265 in patients with MET gene amplifications in blood (circulating tumor DNA)
  Interventions: Drug: MGCD265

INTERVENTIONS:
Drug: MGCD265 — MGCD265 is a small molecule multi-targeted receptor tyrosine kinase inhibitor

SUMMARY:
MGCD265 is an orally administered receptor tyrosine kinase inhibitor that targets MET and other receptors. This study is a Phase 2 trial of MGCD265 in patients with locally advanced, unresectable or metastatic non-small cell lung cancer (NSCLC) that has activating genetic changes of the MET gene (mutation or amplification [increase number of gene copies]). Testing for tumor gene changes can be performed in tumor tissue or blood samples. Patients must have previously received treatment with chemotherapy. The number of patients to be enrolled will depend on how many enrolled patients experience tumor size reduction. MGCD265 will be administered orally, twice daily. The study is designed to evaluate whether the number of patients experiencing tumor size reduction is substantially higher than would be expected with other available treatments.

DETAILED DESCRIPTION:
If testing has not already been performed, the study will provide for the testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-small cell lung cancer
* Metastatic or locally advanced disease
* Prior platinum chemotherapy or immunotherapy
* Test result showing genetic change in MET tumor gene
* At least one tumor that can be measured on a radiographic scan

Exclusion Criteria:

* Prior treatment with inhibitor of MET or HGF
* Prior positive test for EGFR mutation or ALK gene rearrangement
* Uncontrolled tumor in the brain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-10; Primary Completion 2018-04-30 (Actual); Study Completion 2019-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (47):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Clearview Cancer Institute, Huntsville, Alabama
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Providence Saint Joseph Medical Center, Burbank, California
  - Saint Joseph Heritage Healthcare, Fullerton, California
  - University of California San Diego, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of California, San Francisco, San Francisco, California
  - Innovative Clinical Reseach Institute, Whittier, California
  - St. Mary's Regional Cancer Center, Grand Junction, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital - Eugene M. & Christine E. Lynn Cancer Institute, Boca Raton, Florida
  - Sylvester Comprehensive Cancer Center, Deerfield Beach, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Robert H. Lurie Comprehensive Cancer Center of Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Mercy Cancer Center, Mason City, Iowa
  - Oncology-Hematology Associates, PA, Danville, Kentucky
  - Lexington Oncology Associates, LLC, Lexington, Kentucky
  - Kentuckyone Health Cancer and Blood Speacialists, Louisville, Kentucky
  - Christus Saint Frances Cabrini Hospital, Alexandria, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Queens Cancer Center, Jamaica, New York
  - Clinical Research Alliance, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Guthrie Cancer Center, Sayre, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Mary Crowley Cancer Research Centers, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (10):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Saint George Hospital, Kogarah, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Cancer Centre, Clayton, Victoria
  - Austin Health, Heidelberg, Victoria
  - Flinders Medical Centre, Bedford Park
  - Monash Health, Clayton
  - The Tweed Hospital, Tweed Heads
  - Princess Alexandra Hospital, Woolloongabba
- McGill University Health Centre, Montreal, Canada
- Hungary (4):
  - Szent Borbála Kórház, Tatabánya, Komárom-Esztergom
  - Országos Korányi TBC és Pulmonológiai Intézet, Budapest
  - Országos Onkológiai Intézet, Budapest
  - Semmelweis Egyetem, Budapest
- Italy (8):
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Unico Versilia, Lucca
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Europeo di Oncologia Milano, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Unità Sanitaria Locale di Piacenza-Ospedale Guglielmo da Saliceto, Piacenza
  - Azienda Unita Sanitaria Locale di Ravenna, Ravenna
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Torino
- Poland (3):
  - Med Polonia Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Samodzielny Publiczny Zespól Gruzlicy i Chorób Pluc w Olsztynie, Olsztyn, Warmian-Masurian Voivodeship
- South Korea (11):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Saint Vincent Hospital, Suwon, Gyeonggi-do
  - The Catholic University of Korea Saint Vincent's Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Keimyung University Dongsan Medical Center, Daegu
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Veterans Health Service Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Taiwan (6):
  - National Cheng Kung University, Tainan, Tainan CITY
  - Chi Mei Hospital Liouying, Tainan, Tainan
  - Hualien Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - North Bristol NHS Trust, Westbury on Trym, Bristol, England
  - University College London Hospitals NHS Foundation Trust, London, England
  - East and North Hertordshire NHS Trust, Northwood, England
  - Royal Free London NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hong DS, Cappuzzo F, Chul Cho B, Dowlati A, Hussein M, Kim DW, Percent I, Christensen JG, Morin J, Potvin D, Faltaos D, Tassell V, Der-Torossian H, Chao R. Phase II study investigating the efficacy and safety of glesatinib (MGCD265) in patients with advanced NSCLC containing MET activating alterations. Lung Cancer. 2024 Apr;190:107512. doi: 10.1016/j.lungcan.2024.107512. Epub 2024 Feb 22. PMID 38417277
- [Derived] Kollmannsberger C, Hurwitz H, Bazhenova L, Cho BC, Hong D, Park K, Reckamp KL, Sharma S, Der-Torossian H, Christensen JG, Faltaos D, Potvin D, Tassell V, Chao R, Shapiro GI. Phase I Study Evaluating Glesatinib (MGCD265), An Inhibitor of MET and AXL, in Patients with Non-small Cell Lung Cancer and Other Advanced Solid Tumors. Target Oncol. 2023 Jan;18(1):105-118. doi: 10.1007/s11523-022-00931-9. Epub 2022 Dec 2. PMID 36459255

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sponsor approval of each potential patient's genetic testing following prescreening, whether performed by the study central lab or a Sponsor-approved local lab, was filed prior to proceeding to full clinical screening. All patients considered eligible for the study following clinical screening were submitted to Sponsor for registration approval.
Groups:
- MET Activating Mutations in Tumor Tissue: MGCD265 (750 mg BID spray dried dispersion tablet or 1050 mg BID soft-gel capsule) in patients with MET activating mutations in tumor tissue.
- MET Gene Amplifications in Tumor Tissue: MGCD265 (750 mg BID spray dried dispersion tablet or 1050 mg BID soft-gel capsule) in patients with MET gene amplifications in tumor tissue.
- MET Activating Mutations in ctDNA: MGCD265 (750 mg BID spray dried dispersion tablet or 1050 mg BID soft-gel capsule) in patients with MET activating mutations in the blood (circulating tumor DNA).
- MET Gene Amplifications in ctDNA: MGCD265 (750 mg BID spray dried dispersion tablet or 1050 mg BID soft-gel capsule) in patients with MET gene amplifications in the blood (circulating tumor DNA).
Period: Treatment Period
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Started | 28 | 20 | 8 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 28 | 20 | 8 | 12
Not completed — Patient Still on Treatment/Study | 0 | 1 | 1 | 0
Not completed — Adverse Event | 7 | 4 | 0 | 5
Not completed — Lack of Efficacy | 17 | 11 | 5 | 5
Not completed — Global Deterioration of Health | 3 | 3 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Non-compliance | 0 | 0 | 1 | 0
Not completed — Clinical Disease Progression | 0 | 0 | 0 | 1
Period: Survival Follow-up Period
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Started (2 patients on treatment at the time of primary report date) | 28 | 19 | 7 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 28 | 19 | 7 | 12
Not completed — Death | 12 | 14 | 3 | 9
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0 | 1 | 0
Not completed — Study Terminated by Sponsor | 12 | 4 | 2 | 3

BASELINE CHARACTERISTICS:
Population: These figures are based on the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA | Total
Number analyzed (Participants) | 28 | 20 | 8 | 12 | 68
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean (STD) | 70.7 (6.02) | 61.8 (13.17) | 59.1 (7.70) | 64.8 (11.09) | 65.7 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 4 | 6 | 6 | 32
  Male | 12 | 16 | 2 | 6 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 28 | 20 | 7 | 12 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 6 | 2 | 2 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 21 | 13 | 6 | 10 | 50
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 21 | 13 | 6 | 10 | 50
  Black or African American | 2 | 1 | 0 | 0 | 3
  Asian | 4 | 6 | 2 | 2 | 14
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Other | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 2 | 6 | 0 | 2 | 10
  Hungary | 0 | 1 | 0 | 0 | 1
  United States | 23 | 10 | 5 | 7 | 45
  Poland | 0 | 0 | 1 | 2 | 3
  Italy | 0 | 1 | 0 | 1 | 2
  United Kingdom | 1 | 0 | 2 | 0 | 3
  Australia | 2 | 2 | 0 | 0 | 4
Height [Mean (Standard Deviation); unit: cm] — Population: Some patients did not have height recorded at baseline
  cm
    number analyzed (Participants) | 26 | 20 | 4 | 12 | 62
    (all) | 168.63 (9.74) | 173.18 (8.77) | 161.11 (8.10) | 167.70 (8.98) | 169.43 (9.52)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI unable to be calculated in patients with no height recorded at baseline
  kg/m^2
    number analyzed (Participants) | 26 | 20 | 4 | 12 | 62
    (all) | 25.16 (4.58) | 24.92 (4.46) | 22.24 (2.34) | 21.80 (4.18) | 24.24 (4.49)
Weight [Mean (Standard Deviation); unit: kg] | 70.85 (17.64) | 75.33 (17.77) | 60.97 (8.68) | 61.58 (13.56) | 69.37 (16.85)
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self care. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 10 | 6 | 2 | 2 | 20
    1 | 16 | 12 | 6 | 6 | 40
    2 | 2 | 2 | 0 | 4 | 8
    3 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0
Primary Disease Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 22 | 18 | 7 | 6 | 53
  Squamous Cell Carcinoma | 3 | 2 | 1 | 2 | 8
  Large Cell Carcinoma | 0 | 0 | 0 | 2 | 2
  Other | 3 | 0 | 0 | 2 | 5
Current Stage [Count of Participants; unit: Participants]
  Locally Advanced | 1 | 1 | 0 | 1 | 3
  Metastatic | 27 | 19 | 8 | 11 | 65
Smoking History [Count of Participants; unit: Participants]
  Lifetime Non-Smoker | 10 | 2 | 3 | 2 | 17
  Current Smoker | 0 | 4 | 1 | 3 | 8
  Past Smoker | 18 | 14 | 4 | 7 | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective disease response is defined as the percent of patients documented by investigator assessment to have a confirmed Complete Response (CR) or Partial Response (PR) in accordance with the Response Evaluation Criteria in Solid Tumors (RECIST 1.1) for target and non-target lesions as assessed by CT or MRI. CR is defined as complete disappearance of all target lesions with the exception of nodal disease; PR is defined as >=30% decrease under baseline of the sum of diameters of all target measurable lesions; Stable Disease (SD) is concluded when the response does not qualify for CR, PR or Progression; Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions.
Time Frame: Up to 3 months
Population: Modified Intent-to-Treat (mITT) Population defined as all patients who received at least one dose of MGCD265
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 28 | 20 | 8 | 12
percentage of participants | 10.7 [2.27 to 28.23] | 15.0 [3.21 to 37.89] | 25.0 [3.19 to 65.09] | 0.0 [0.00 to 26.46]
Statistical Analysis 1: Comparison: MET Activating Mutations in Tumor Tissue; Test type: Superiority — An exact test for single proportion (two-sided a=5%) will be performed to test H0: ORR <=20% against H1: ORR >20%; p = 0.94, exact test; Objective response rate = 10.7, 95% CI 2-sided [2.27 to 28.23]
Statistical Analysis 2: Comparison: MET Gene Amplifications in Tumor Tissue; Test type: Superiority; p = 0.79, exact test; Objective response rate = 15.0, 95% CI 2-sided [3.21 to 37.89]
Statistical Analysis 3: Comparison: MET Activating Mutations in ctDNA; Test type: Superiority; p = 0.47, Exact Test; Objective response rate = 25.0, 95% CI 2-sided [3.19 to 65.09]
Statistical Analysis 4: Comparison: MET Gene Amplifications in ctDNA; Test type: Superiority; p > 0.999, Exact test; Objective response rate = 0, 95% CI 2-sided [0.00 to 26.46]

2. Secondary Outcome: Duration of Response
Description: Duration of Response (DR) will be defined as the time from date of the first documentation of objective tumor response (CR or PR) to the first documentation of Objective Progression of Disease (PD) or to death due to any cause in the absence of documented PD.
Time Frame: From date of the first documentation of objective tumor response (CR or PR) to the first documentation of Objective Progression of Disease (PD) or to death due to any cause in the absence of documented PD, assessed up to 24 months.
Population: Modified Intent-to-Treat (mITT) Population defined as all patients who received at least one dose of MGCD265
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 3 | 3 | 2 | 0
days | 85 [82 to 132] | 170 [120 to 170] | NA [77 to NA] — Median DR and upper bound of 95% CI for median DR are not estimable. Median not reached/small number of events. |

3. Secondary Outcome: Progression Free Survival
Description: Progression-free survival (PFS) will be defined as the time from date of first study treatment to first PD or death due to any cause in the absence of documented PD. Per RECIST 1.1, Progressive Disease (PD) is defined as a 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm, or unequivocal progression of pre-existing non-target lesions.
Time Frame: The time from date of first study treatment to first PD or death due to any cause in the absence of documented PD, up to 24 months.
Population: Modified Intent-to-Treat (mITT) Population defined as all patients who received at least one dose of MGCD265
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 28 | 20 | 8 | 12
months | 3.95 [2.11 to 4.18] | 4.84 [1.35 to 5.53] | 3.39 [1.28 to NA] — Upper bound of 95% CI for median PFS is not estimable due to small number of events. | 2.76 [1.48 to 4.01]

4. Secondary Outcome: 1-Year Survival Rate
Description: 1-Year Survival will be defined as the probability of survival at 1 year after the first dose.
Time Frame: From date of first study treatment to death due to any cause, assessed up to 12 months
Population: Modified Intent-to-Treat (mITT) Population defined as all patients who received at least one dose of MGCD265
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 28 | 20 | 8 | 12
percentage | 50.47 [27.49 to 69.62] | 34.92 [14.05 to 56.89] | 54.69 [13.72 to 83.24] | 13.89 [0.86 to 44.05]

5. Secondary Outcome: Overall Survival
Description: Overall Survival will be defined as the time from date of first study treatment to death due to any cause
Time Frame: From date of first study treatment to death due to any cause, assessed up to 24 months.
Population: Modified Intent-to-Treat (mITT) Population defined as all patients who received at least one dose of MGCD265
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 28 | 20 | 8 | 12
months | 16.32 [4.01 to NA] — Upper bound of 95% CI for median OS is not estimable due to small number of events. | 7.04 [1.84 to 14.93] | NA [.89 to NA] — Median OS and upper bound of 95% CI for median OS are not estimable. Median not reached/small number of events. | 4.08 [1.22 to 11.05]

6. Secondary Outcome: Number of Patients Experiencing Treatment-emergent Adverse Events
Description: Number of patients experiencing treatment-emergent adverse events.
Time Frame: Date of first dose to 28 days after the last dose, up to an average of 5.1 months on treatment.
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 28 | 20 | 8 | 12
Participants | 28 | 20 | 8 | 12

7. Secondary Outcome: Blood Plasma Concentration of MGCD265 - AUC0-6
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose.
Population: PK Analysis Set consisted of all patients who received at least one dose of active study drug and had sufficient data to assess any of the PK parameters.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Groups:
- Tablet 750 mg BID C1D1: Tablet formulation, 750 mg, BID, Cycle 1 Day 1
- Tablet 750 mg BID C1D15: Tablet formulation, 750 mg, BID, Cycle 1 Day 15
- Soft Gel 1050 mg BID C1D1: Soft Gel formulation, 1050 mg, BID, Cycle 1 Day 1
- Soft Gel 1050 mg BID C1D15: Soft Gel formulation, 1050 mg, BID, Cycle 1 Day 15
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15
Number analyzed (Participants) | 46 | 30 | 17 | 13
h*ng/mL | 250.8 (98.0) | 1565 (54.0) | 185.5 (98.8) | 1837 (51.3)

8. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Cmax
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. On Cycle 2, samples were collected on Day 1 and Day 15 at pre-dose and at 6 hours post-dose (4-8 hours). Note: Assessment of Cmax and Tmax are limited by the sparse blood sampling schedule post dose (i.e., only 2 blood draws post-dose in Cycle 1 and only 1 sample collected post-dose in Cycle 2). The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. Cycle 2, Day 1 and Day 15 at pre-dose and at 6 hours post-dose (4-8 hours).
Population: PK Analysis Set consisted of all patients who received at least one dose of active study drug and had sufficient data to assess any of the PK parameters. No results are reported for C2D15 because the number of observations were less than 3 for the 1050 mg BID (Soft Gel Capsule).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Tablet 750 mg BID C2D1: Tablet formulation, 750 mg, BID, Cycle 2 Day 1
- Tablet 750 mg BID C2D15: Tablet formulation, 750 mg, BID, Cycle 2 Day 15
- Soft Gel 1050 mg BID C2D1: Soft Gel formulation, 1050 mg, BID, Cycle 2 Day 1
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15 | Tablet 750 mg BID C2D1 | Tablet 750 mg BID C2D15 | Soft Gel 1050 mg BID C2D1
Number analyzed (Participants) | 46 | 30 | 17 | 13 | 29 | 5 | 3
ng/mL | 69.77 (87.1) | 279.2 (54.6) | 60.49 (103.9) | 328.1 (49.8) | 214 (69.4) | 138 (100.0) | 386 (13.9)

9. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Ctrough
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. On Cycle 2, samples were collected on Day 1 and Day 15 at pre-dose and at 6 hours post-dose (4-8 hours). The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15 | Tablet 750 mg BID C2D1 | Tablet 750 mg BID C2D15 | Soft Gel 1050 mg BID C2D1
Number analyzed (Participants) | 0 | 36 | 0 | 15 | 35 | 5 | 8
ng/mL |  | 264 (52.5) |  | 337 (59.2) | 203 (80.9) | 255 (37.5) | 345 (48.5)

10. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Accumulation Ratio AUC0-6
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose. Accumulation Ratio AUC0-6 = AUC0-6 C1D15/ AUC0-6 C1D1.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15
Number analyzed (Participants) | 0 | 30 | 0 | 13
ratio |  | 6.42 (87.2) |  | 9.88 (96.4)

11. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Accumulation Ratio Cmax
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose. Accumulation Ration Cmax = Cmax C1D15/ Cmax C1D1.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15
Number analyzed (Participants) | 0 | 30 | 0 | 13
ratio |  | 4.07 (79.7) |  | 5.35 (100.9)

12. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Peak to Trough Ratio
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose. Peak to trough ratio calculated as C1D15 Cmax/Ctrough.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose.
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15
Number analyzed (Participants) | 0 | 30 | 0 | 13
ratio |  | 1.09 (13.4) |  | 1.08 (10.4)

13. Secondary Outcome: Blood Plasma Concentration of MGCD265 - Tmax
Description: Blood samples for PK assessment were to be taken on Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose. Note: Assessment of Cmax and Tmax are limited by the sparse blood sampling schedule post dose (i.e., only 2 blood draws post-dose in Cycle 1 and only 1 sample collected post-dose in Cycle 2). The number of patients reported for each PK parameter was dependent on the actual number of blood samples collected post-dose.
Time Frame: Cycle 1, Day 1 and Day 15 at pre-dose and at 2 hours (1-3 hours) and 6 hours (4-8 hours) post-dose.
Population: as for outcome 7
Measure: Median (Full Range); unit: hours
Arm/Group | Tablet 750 mg BID C1D1 | Tablet 750 mg BID C1D15 | Soft Gel 1050 mg BID C1D1 | Soft Gel 1050 mg BID C1D15
Number analyzed (Participants) | 46 | 30 | 17 | 13
hours | 6.00 [2.00 to 6.00] | 2.00 [2.00 to 6.00] | 6.00 [6.00 to 6.00] | 6.00 [2.00 to 6.00]

14. Secondary Outcome: Assess Correlation Between Selected Tumor Gene Alterations Using Different Analytical Techniques in Tumor Tissue and Circulating Tumor Deoxyribonucleic Acid (ctDNA) - MET Activating Mutations
Description: Only a sub-set of patients had different molecular techniques completed, therefore a correlation analysis was not performed. Patients with positive identification by two different analytical techniques are tabulated for MET Activating Mutations.
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Groups:
- MET Activating Mutations: Patients with MET Activating Mutations
Arm/Group | MET Activating Mutations
Number analyzed (Participants) | 11
Participants
  Positive by both PCR and NGS | 9
  Positive by PCR and Negative by NGS | 1
  Negative by PCR and Positive by NGS | 1
  Negative by both PCR and NGS | 0

15. Secondary Outcome: Assess Correlation Between Selected Tumor Gene Alterations Using Different Analytical Techniques in Tumor Tissue and Circulating Tumor Deoxyribonucleic Acid (ctDNA) - MET Gene Amplifications
Description: Only a sub-set of patients had different molecular techniques completed, therefore a correlation analysis was not performed. Patients with positive identification by two different analytical techniques are tabulated for MET Gene Amplifications.
Time Frame: At baseline
Measure: Count of Participants; unit: Participants
Groups:
- MET Gene Amplifications: Patients with MET Gene Amplifications
Arm/Group | MET Gene Amplifications
Number analyzed (Participants) | 21
Participants
  Positive by both FISH and NGS | 8
  Positive by FISH and Negative by NGS | 6
  Negative by FISH and Positive by NGS | 7
  Negative by both FISH and NGS | 0

16. Secondary Outcome: Assess Change in Genetic Alteration Status in ctDNA With MGCD265 Treatment Over Time in the Selected Population
Time Frame: At baseline and at time of confirmation of response to treatment
Population: The study was closed early due to sponsor portfolio prioritization and not due to any patient safety issues. Based on limited individual patient data for whom baseline and post-treatment values were available, the statistical analyses as planned could not be performed. Screening and end of treatment detection results provided.
Measure: Number; unit: participants
Groups:
- MET Activating Mutation: MET Exon 14 deletion mutation
- MET Gene Amplification: MET activating mutation
Arm/Group | MET Activating Mutation | MET Gene Amplification
Number analyzed (Participants) | 2 | 2
participants
  Detected at Screening | 2 | 2
  Detected at End of Treatment | 2 | 1

17. Secondary Outcome: Blood Plasma Concentration of Soluble MET (sMET) Biomarker
Description: MET Activating Mutations in ctDNA. Change from Baseline - Cycle 2 Day 15 - Pre-Dose Standard Deviation not evaluable
Time Frame: Cycle 1 and Cycle 2
Population: The Pharmacodynamics Evaluable Population Population defined as all patients in the mITT population for whom PD analytical results were available. Overall number of participants analyzed at baseline and post-baseline are different due to samples not being collected post-baseline for some patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA
Number analyzed (Participants) | 22 | 17 | 4 | 9
pg/mL
  Baseline | 443494.7 (228345.48) | 461985.2 (122069.25) | 450112.5 (80809.29) | 961383.1 (1665608.92)
  Actual - Cycle 1 Day 15 - Pre-Dose: number analyzed (Participants) | 20 | 15 | 4 | 8
  Actual - Cycle 1 Day 15 - Pre-Dose | 577631.4 (221350.47) | 568938.8 (129859.54) | 594277.3 (49746.18) | 775242.8 (679349.02)
  Change from Baseline - Cycle 1 Day 15 - Pre-Dose: number analyzed (Participants) | 19 | 15 | 4 | 8
  Change from Baseline - Cycle 1 Day 15 - Pre-Dose | 122074.7 (166978.07) | 94110.4 (87158.09) | 144164.8 (51740.94) | -257537.5 (1102955.10)
  Actual - Cycle 2 Day 1 - Pre-Dose: number analyzed (Participants) | 20 | 17 | 4 | 9
  Actual - Cycle 2 Day 1 - Pre-Dose | 560790.3 (216802.34) | 582800.9 (140742.66) | 662385.3 (41039.78) | 742344.9 (620417.99)
  Change from Baseline - Cycle 2 Day 1 - Pre-Dose: number analyzed (Participants) | 19 | 17 | 4 | 9
  Change from Baseline - Cycle 2 Day 1 - Pre-Dose | 144802.6 (158943.04) | 120815.6 (133979.33) | 212272.8 (86344.15) | -219038.2 (1085522.39)
  Actual - Cycle 2 Day 15 - Pre-Dose: number analyzed (Participants) | 14 | 11 | 1 | 5
  Actual - Cycle 2 Day 15 - Pre-Dose | 551625.9 (234249.28) | 630505.5 (133180.58) | 482109.0 | 628011.8 (291532.85)
  Change from Baseline - Cycle 2 Day 15 - Pre-Dose: number analyzed (Participants) | 13 | 11 | 1 | 5
  Change from Baseline - Cycle 2 Day 15 - Pre-Dose | 96641.3 (144021.14) | 169374.6 (70996.25) | 44093.0 | 184161.0 (161224.04)

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: All Cause Mortality includes deaths that occurred in the Treatment Period and the Survival Follow-Up Period.
Groups:
- Total: All patients
Arm/Group | MET Activating Mutations in Tumor Tissue | MET Gene Amplifications in Tumor Tissue | MET Activating Mutations in ctDNA | MET Gene Amplifications in ctDNA | Total
All-Cause Mortality (participants affected / at risk) | 12/28 | 14/20 | 3/8 | 9/12 | 38/68
Serious Adverse Events (participants affected / at risk) | 12/28 | 10/20 | 4/8 | 7/12 | 33/68
Other Adverse Events (participants affected / at risk) | 28/28 | 20/20 | 7/8 | 12/12 | 67/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MET Activating Mutations in Tumor Tissue (N=28) | MET Gene Amplifications in Tumor Tissue (N=20) | MET Activating Mutations in ctDNA (N=8) | MET Gene Amplifications in ctDNA (N=12) | Total (N=68)
Myocardial Infarction (Cardiac disorders) | 2 | 0 | 0 | 0 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0 | 1
Hepatic haemorrhage (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 3 | 1 | 0 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 0 | 3 | 6
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5 | 1 | 4 | 15
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MET Activating Mutations in Tumor Tissue (N=28) | MET Gene Amplifications in Tumor Tissue (N=20) | MET Activating Mutations in ctDNA (N=8) | MET Gene Amplifications in ctDNA (N=12) | Total (N=68)
Anaemia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 1 | 6
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 1 | 1 | 0 | 3
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1
Eye discharge (Eye disorders) | 0 | 0 | 1 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 1 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 1
Visual impairment (Eye disorders) | 2 | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 1 | 4 | 12
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 5
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 3 | 10
Diarrhoea (Gastrointestinal disorders) | 22 | 18 | 7 | 10 | 57
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 4
Flatulence (Gastrointestinal disorders) | 5 | 1 | 0 | 1 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 3
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 15 | 9 | 6 | 6 | 36
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 7 | 8 | 6 | 6 | 27
Asthenia (General disorders) | 2 | 3 | 1 | 1 | 7
Catheter site pain (General disorders) | 0 | 1 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 0 | 1 | 3
Face oedema (General disorders) | 1 | 0 | 2 | 0 | 3
Fatigue (General disorders) | 13 | 8 | 5 | 7 | 33
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0 | 2
Malaise (General disorders) | 2 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 1 | 3
Oedema (General disorders) | 2 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 8 | 5 | 3 | 0 | 16
Pain (General disorders) | 1 | 3 | 0 | 0 | 4
Peripheral swelling (General disorders) | 2 | 1 | 0 | 1 | 4
Pyrexia (General disorders) | 1 | 0 | 1 | 0 | 2
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1
Perforation bile duct (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Mucosal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 1 | 1 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 3 | 1 | 0 | 0 | 4
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 2
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 14 | 8 | 3 | 5 | 30
Aspartate aminotransferase increased (Investigations) | 12 | 9 | 3 | 4 | 28
Blood creatine increased (Investigations) | 0 | 0 | 1 | 0 | 1
Blood alkaline phosphatase (Investigations) | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 3 | 2 | 0 | 8
Blood lactate dehydrogenase increased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 1 | 0 | 1 | 0 | 2
Capillary nail refill test abnormal (Investigations) | 0 | 1 | 0 | 0 | 1
Haemoglobin (Investigations) | 0 | 0 | 0 | 1 | 1
Inflammatory marker increased (Investigations) | 0 | 1 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 1 | 0 | 0 | 4
Platelet count decreased (Investigations) | 3 | 2 | 0 | 1 | 6
Platelet count increased (Investigations) | 0 | 0 | 1 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 1 | 2
Weight decreased (Investigations) | 4 | 0 | 0 | 0 | 4
Weight increased (Investigations) | 1 | 1 | 0 | 0 | 2
White blood cell count decreased (Investigations) | 2 | 0 | 1 | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 12 | 6 | 3 | 4 | 25
Dehydration (Metabolism and nutrition disorders) | 6 | 2 | 0 | 1 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 3 | 10
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 1 | 1 | 2 | 7
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 1 | 2 | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 4 | 2 | 2 | 17
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 5 | 2 | 0 | 0 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 0 | 4
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 1 | 10
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 4
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 2
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 4 | 3 | 3 | 0 | 10
Dysgeusia (Nervous system disorders) | 2 | 1 | 2 | 0 | 5
Headache (Nervous system disorders) | 4 | 2 | 0 | 0 | 6
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 2 | 0 | 0 | 1 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 1 | 0 | 0 | 3
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Dysphemia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 2
Oliguria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 3 | 1 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8 | 2 | 4 | 20
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3 | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 2 | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 4
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 0 | 1 | 8
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 2
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0 | 0 | 2
Hypotension (Vascular disorders) | 3 | 0 | 0 | 0 | 3
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Early closure of the study is due to sponsor portfolio prioritization and not due to any patient safety issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can not disclose, discuss, or publish study results until final manuscript has been published.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-23): https://cdn.clinicaltrials.gov/large-docs/33/NCT02544633/Prot_SAP_000.pdf